CLINICAL TRIAL: NCT06072690
Title: The Impact of Dual Bronchodilation on Respiratory and Cardiovascular Systems in Patients With Newly Diagnosed Moderate-to-severe Chronic Obstructive Pulmonary Disease
Brief Title: Respiratory and Cardiovascular Alterations in Patients With Chronic Obstructive Pulmonary Disease
Status: Recruiting | Type: Observational
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Skaidrius Miliauskas, Head of Pulmonology Department, Professor, Lithuanian University of Health Sciences
Other Study IDs: COPDCVS1
Record Dates: First submitted 2023-09-27; First posted 2023-10-10 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Chronic Obstructive Pulmonary Disease Moderate; Chronic Obstructive Pulmonary Disease Severe; Cardiovascular Diseases; Quality of Life
Keywords: COPD; cardiac autonomic integrity; cardiac function; dual bronchodilation; biomarkers; quality of life
MeSH Terms: conditions — Cardiovascular Diseases; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COPD group: Patients of any gender aged 40 years and older with newly diagnosed treatment-naive moderate-to-severe chronic obstructive pulmonary disease will have a comprehensive cardiovascular and respiratory examination as well as evaluation of quality of life before the treatment and after 12 weeks of treatment with dual bronchodilation.
- Non-COPD group: Subjects 40 years and older without respiratory conditions with similar age, gender and cardiovascular comorbidity profile

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a major cause of disability and death worldwide. People with COPD often have cardiovascular diseases (CVDs) that are associated with increased risk for hospitalization and prolonged stay as well as all-cause and CVD-related mortality. Nevertheless, CVDs in patients with COPD are tend to be underestimated in clinical practice. Mechanisms that define the relation between COPD and cardiovascular morbidity include lung hyperinflation, hypoxia, pulmonary hypertension, systemic inflammation and oxidative stress, exacerbation, shared risk factors and COPD phenotypes. Recently, some authors have announced that COPD treatment with dual bronchodilation may not only improve pulmonary function and quality of life, but also have a positive effect on cardiac function in cardiac magnetic resonance imaging (MRI) or two-dimensional cardiac ultrasound for the assessments. The aim of this study is to specify the state of respiratory and cardiovascular systems as well as exercise capacity and quality of life in patients with newly diagnosed moderate-to-severe COPD and to evaluate their changes after short-term treatment with dual bronchodilation. We hypothesize that patients with newly diagnosed COPD and no previous records of cardiac diseases and no apparent signs of heart failure have significantly impaired cardiac autonomic integrity that precedes to increased risk of cardiovascular events. It is believed that cardiac autonomic integrity might significantly improve with dual bronchodilation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Aged 40 years and older
* Smoking index of 10 pack-years and more
* Newly diagnosed chronic obstructive pulmonary disease (COPD) with forced expiratory volume in 1 second (FEV1) 30-79 percent of predicted and forced expiratory volume in 1 second to forced vital capacity ratio (FEV1/FVC) less than 70 percent of predicted.

Exclusion Criteria:

* Active lung infection
* Present or previously treated lung cancer
* Alpha-1 antitrypsin deficiency
* Diagnosed interstitial lung disease
* Previously diagnosed asthma
* Diagnosed chronic hypercapnic respiratory failure
* Treatment with systemic glucocorticoids
* Unstable ischaemic heart disease
* Pregnancy
* Present cardiac arrhythmias
* Uncontrolled arterial hypertension
* Dementia and other mental states that determine patient's inability to consent
* Other medical conditions that in the opinion of the investigator disqualify the subject for inclusion

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The cohort will be selected from patients with clinical signs of COPD reffered to the tertiary care outpatient clinic by general physicians from the primary and secondary care clinics.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in cardiopulmonary exercise testing at week 12 | Baseline and week 12
  The effect of dual bronchodilation on cardiopulmonary exercise test results in patients with newly diagnosed moderate-to-severe chronic obstructive pulmonary disease
Change from baseline in health-related quality of life at week 12 | Baseline and week 12
  The effect of dual bronchodilation on health related quality of life (evaluating using the Short Form 36 Health Survey (SF-36) Questionnaire) in patients with newly diagnosed moderate-to-severe chronic obstructive pulmonary disease

SECONDARY OUTCOMES:
Change from baseline in forced expiratory volume in 1 second at week 12 | Baseline and week 12
  The effect of dual bronchodilation on forced expiratory volume in 1 second (FEV1) in patients with newly diagnosed moderate-to-severe chronic obstructive pulmonary disease
Change from baseline in forced vital capacity at week 12 | Baseline and week 12
  The effect of dual bronchodilation on forced vital capacity (FVC) in patients with newly diagnosed moderate-to-severe chronic obstructive pulmonary disease
Change from baseline in diffusing capacity of the lungs for carbon monoxide at week 12 | Baseline and week 12
  The effect of dual bronchodilation on diffusing capacity of the lungs for carbon monoxide (DLCO) in patients with newly diagnosed moderate-to-severe chronic obstructive pulmonary disease
Change from baseline in residual volume at week 12 | Baseline and week 12
  The effect of dual bronchodilation on residual volume (RV) in patients with newly diagnosed moderate-to-severe chronic obstructive pulmonary disease
Change from baseline in residual volume to total lung capacity ratio at week 12 | Baseline and week 12
  The effect of dual bronchodilation on residual volume to total lung capacity ratio (RV/TLC) in patients with newly diagnosed moderate-to-severe chronic obstructive pulmonary disease
Change from baseline in forced residual capacity to total lung capacity ratio at week 12 | Baseline and week 12
  The effect of dual bronchodilation on forced residual capacity to total lung capacity ratio (FRC/TLC) in patients with newly diagnosed moderate-to-severe chronic obstructive pulmonary disease
Change from baseline in right ventricle end-systolic volume index at week 12 | Baseline and week 12
  The effect of dual bronchodilation on right ventricle end-systolic volume index (RVESVi) in patients with newly diagnosed moderate-to-severe COPD
Change from baseline in right ventricle end-diastolic volume index at week 12 | Baseline and week 12
  The effect of dual bronchodilation on right ventricle end-diastolic volume index (RVEDVi) in patients with newly diagnosed moderate-to-severe COPD
Change from baseline in on left ventricle end-systolic volume index at week 12 | Baseline and week 12
  The effect of dual bronchodilation on left ventricle end-systolic volume index (LVESVi) in patients with newly diagnosed moderate-to-severe COPD
Change from baseline in left ventricle end-diastolic volume index at week 12 | Baseline and week 12
  The effect of dual bronchodilation on left ventricle end-diastolic volume index (LVEDVi) in patients with newly diagnosed moderate-to-severe COPD
Change from baseline in stroke volume index at week 12 | Baseline and week 12
  The effect of dual bronchodilation on stroke volume index (SVi) in patients with newly diagnosed moderate-to-severe COPD
Change from baseline in right ventricular strains at week 12 | Baseline and week 12
  The effect of dual bronchodilation on right ventricular strains in patients with newly diagnosed moderate-to-severe COPD
Change from baseline in washout rate at week 12 | Baseline and week 12
  The effect of dual bronchodilation on washout rate (WR) in cardiac sympathetic imaging with meta-iodobenzylguanidine in patients with newly diagnosed moderate-to-severe COPD
Change from baseline in heart to mediastinum ratio at week 12 | Baseline and week 12
  The effect of dual bronchodilation on early and late heart to mediastinum ratio (HMR) in cardiac sympathetic imaging with meta-iodobenzylguanidine in patients with newly diagnosed moderate-to-severe COPD
Change from baseline in left ventricle total defect score at week 12 | Baseline and week 12
  The effect of dual bronchodilation on early and late left ventricle early total defect score (TDS) in cardiac sympathetic imaging with meta-iodobenzylguanidine in patients with newly diagnosed moderate-to-severe COPD
Differences in health-related quality of life between COPD and non-COPD individuals | Baseline
Differences in exercise capacity between COPD and non-COPD individuals | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Skaidrius Miliauskas, PhD, Prof., Principal Investigator — Lithuanian University of Health Sciences, Medical Academy, Department of Pulmonology
Locations (1):
- Lithuanian University of Health Sciences, Kaunas, Lithuania